CLINICAL TRIAL: NCT00633243
Title: Effective Treatment of Hepatitis C in Substance Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, R. Douglas Bruce, MD, MA, Assistant Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0702002306; NIDA 022143
Record Dates: First submitted 2008-02-29; First posted 2008-03-11 (Estimated); Results first posted 2012-11-20 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Hepatitis C; Opiate Dependence
MeSH Terms: conditions — Hepatitis C; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified Directly Observed Therapy (mDOT) (Experimental): Hepatitis C Virus (HCV) Treatment in Modified Directly Observed Therapy (mDOT) in Methadone Maintenance Treatment (MMT)
  Interventions: Procedure: Modified Directly Observed Therapy (mDOT)
- Self-Administered Therapy at Liver Specialty Clinic (SAT) (Active Comparator): Hepatitis C virus (HCV) at a liver specialty clinic as self-administered therapy
  Interventions: Procedure: Self-Administered Therapy (SAT)

INTERVENTIONS:
Procedure: Modified Directly Observed Therapy (mDOT)
  Arms: Modified Directly Observed Therapy (mDOT)
Procedure: Self-Administered Therapy (SAT)
  Arms: Self-Administered Therapy at Liver Specialty Clinic (SAT)

SUMMARY:
We hypothesize that integrating Hepatitis C into methadone and buprenorphine treatment will improve Hepatitis C outcomes as well as drug treatment outcomes in patients who are addicted to opiates. We will test this hypothesis by randomly assigning patients to receive integrated or separated care. The first group will receive Hepatitis C treatment and substance abuse treatment contemporaneously at the South Central Rehabilitation Center (SCRC). They will take both methadone or buprenorphine and Hepatitis C medications under the daily (methadone) or weekly (buprenorphine) observation of a health care provider. The second group will receive substance abuse treatment at SCRC, and go to another facility to receive Hepatitis C treatment services. These participants will take their medications on their own (without observation).

We will look at outcomes such as Hepatitis C viral loads, adherence to medications, and drug treatment outcomes such as receipt of buprenorphine and methadone and urine toxicology testing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a DSM IV diagnosis of opioid dependence who are currently enrolled in methadone or buprenorphine maintenance at South Central Rehabilitation Center in good standing (opiate free urine with positive methadone or buprenorphine, respectively) for at least 30 days.
* Hepatitis C infection as evidenced by a positive HCV antibody and a detectable HCV RNA.

Exclusion Criteria:

* Suicidal or homicidal ideation
* Psychiatric condition that is not stable
* Pregnancy (RBV is a Class C drug during pregnancy)
* Pending court case or warrant which would interrupt treatment
* Decompensated cirrhosis (Child's Class B or C) or presence of hepatocellular carcinoma
* HIV+ with CD4<200 or CD4>200 and VL>5,000 copies/mL
* Platelet count < 75,000 /mL
* Hemoglobin < 10 mg/dL
* Absolute neutrophil count <1500 cells/mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Douglas Bruce, M.D., Principal Investigator — Yale University
Locations (1):
- South Central Rehabilitation Agency, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited over a 3-year period (2007-2010) from a substance abuse treatment clinic in New Haven, CT. Those with evidence of infection with HCV were subsequently seen by a medical provider to evaluate for HCV treatment, and if found to be appropriate, were referred to the research assistant.
Pre-assignment Details: Subjects were eligible for participation if they were prescribed methadone and were opioid negative in the past 30 days, age 18 years or older, underwent documented HIV testing, competent to provide informed consent, had stable mental health status, and met the following criteria for HCV treatment: detectable HCV RNA and genotype testing.
Groups:
- Modified Directly Observed Therapy (mDOT): Subjects received modified directly observed therapy (mDOT) as part of an adherence intervention. Clinical nurses administered all methadone doses and co-administered the morning weight-based ribavirin (RBV) dose. The evening dose of RBV was prepackaged by a pharmacist accessible for the subject to self-administer 12 hours later. Pegylated interferon alfa-2a(PEG) was administered to mDOT subjects weekly by a licensed practitioners. All mDOT subjects who earned take-home bottles for methadone also received take-home doses of RBV.
- Self-Administered Therapy (SAT): Subjects received their methadone remote from their site of HCV treatment. HCV treatment was provided within the Yale Liver Center, the university-based liver specialty clinic. All subjects in this arm were taught how to self-administer therapy (SAT), the pegylated interferon alfa-a (PEG) and weight-based ribavirin (RBV). Subjects followed a pre-specified time period of attending the Liver Center for clinical follow-up and blood work.
Period: Overall Study
Arm/Group | Modified Directly Observed Therapy (mDOT) | Self-Administered Therapy (SAT)
Started | 12 | 9
Completed | 11 | 2
Not Completed | 1 | 7
Not completed — Withdrawal by Subject | 0 | 1
Not completed — incarceration | 0 | 2
Not completed — Homeless--no refrigeration for meds | 0 | 1
Not completed — Not comfortable with self-injecting | 0 | 1
Not completed — Mental Health--Depression | 0 | 1
Not completed — Couldn't tolerate side-effects | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Modified Directly Observed Therapy (mDOT): Subjects received modified directly observed therapy (mDOT) as part of an adherence intervention. Clinical nurses administered all methadone doses and co-administered the morning RBV dose. The evening dose of RBV was prepackaged by a pharmacist accessible for the subject to self-administer 12 hours later. PEG was administered to mDOT subjects weekly by a licensed practitioners. All mDOT subjects who earned take-home bottles for methadone also received take-home doses of RBV.
- Self-Administered Therapy (SAT): Subjects received their methadone remote from their site of HCV treatment. HCV treatment was provided within the Yale Liver Center, the university-based liver specialty clinic. All subjects in this arm were taught how to self-administer therapy (SAT), the PEG and RBV. Subjects followed a pre-specified time period of attending the Liver Center for clinical follow-up and blood work.
- Total: Total of all reporting groups
Arm/Group | Modified Directly Observed Therapy (mDOT) | Self-Administered Therapy (SAT) | Total
Number analyzed (Participants) | 12 | 9 | 21
Age Continuous [Mean (Full Range); unit: years] | 40 [29 to 51] | 43 [36 to 54] | 42 [29 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Sustained Virologic Response (SVR)
Description: SVR is defined as continued undetectable HCV viral load at 24 weeks
Time Frame: 24 weeks (end of treatment)
Population: All subjects in mDOT arm and SAT arm who completed treatment.
Measure: Number; unit: participants
Arm/Group | Modified Directly Observed Therapy (mDOT) | Self-Administered Therapy (SAT)
Number analyzed (Participants) | 12 | 4
participants | 7 | 1

ADVERSE EVENTS:
Arm/Group | Modified Directly Observed Therapy (mDOT) | Self-Administered Therapy (SAT)
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9

LIMITATIONS AND CAVEATS:
This trial contains a small sample size of patients with considerable comorbidity and is drawn from one specialized treatment setting. Our conclusions will need empiric testing within carefully conducted RCTs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No